CLINICAL TRIAL: NCT07316049
Title: Construction and Evaluation of an Intelligent Decision System for Reperfusion Therapy in Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LingBao
Record Dates: First submitted 2025-12-02; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-10

CONDITIONS: Acute Ischemic Stroke
Keywords: Reperfusion Therapy; Artificial Intelligence; Clinical Decision Support System
MeSH Terms: conditions — Ischemic Stroke | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Twenty certified stroke centers will be randomized 1:1 to LingBao-assisted care or standard care.
Who Masked: Outcomes Assessor
Masking Description: This is an open-label cluster trial. Neither participants nor investigators are blinded to group assignment. Outcome assessment at 90 days (mRS) will be performed by trained assessors unaware of treatment allocation when feasible.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LingBao-Assisted Care (Experimental): Participants enrolled at stroke centers assigned to the LingBao-assisted group will receive routine clinical care for acute ischemic stroke, with optional use of the LingBao System (Stroke Reperfusion Intelligent Decision System, SRIDS) as a clinical decision support tool during evaluation and management for reperfusion therapy.
  The LingBao System integrates patient demographic, clinical, and imaging data; automatically estimates onset-to-treatment windows; screens contraindications; and provides guideline-concordant recommendations for intravenous thrombolysis and/or endovascular therapy with evidence grading. All final treatment decisions remain at the discretion of the treating physicians.
  Interventions: Other: LingBao System
- Standard Care (Active Comparator): Participants enrolled at stroke centers assigned to the control group will receive standard care for acute ischemic stroke according to current national and international guidelines.
  Clinicians in these centers will not access or use the LingBao System during the study period. All diagnostic and therapeutic decisions will follow usual institutional practice without AI-based support.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: LingBao System — The LingBao System is an artificial intelligence-enabled clinical decision support platform developed to assist physicians in evaluating and managing patients with acute ischemic stroke (AIS) who are candidates for reperfusion therapy.
  The system integrates routinely available clinical and imaging data, automatically estimates onset-to-treatment windows, screens contraindications, and displays guideline-concordant recommendations for intravenous thrombolysis and/or endovascular therapy along with corresponding evidence levels.
  LingBao is intended for use by trained clinicians as an informational tool within standard care pathways. It does not replace physician judgment, modify treatment protocols, or deliver any direct therapeutic intervention.
  LingBao will be available only at centers randomized to the intervention arm ("LingBao-Assisted Care"). Clinicians at control centers ("Standard Care") will not use the system during the study period.
  Other Names: LingBao AI Decision Platform; SRIDS; Intelligent Stroke Reperfusion Decision Support System
  Arms: LingBao-Assisted Care
Other: Standard Care — Participants at stroke centers assigned to the Standard Care arm will receive routine clinical management for acute ischemic stroke (AIS) according to current national and international guidelines.
  Arms: Standard Care

SUMMARY:
This multicenter, cluster-randomized controlled trial will evaluate the effectiveness and safety of the LingBao System, an AI-enabled clinical decision support platform for reperfusion therapy in acute ischemic stroke (AIS). Twenty certified stroke centers will be randomized 1:1 to LingBao-assisted care or standard care. Consecutive patients aged 18 years or older who present within 24 hours of symptom onset or last-known-well and are evaluated for intravenous thrombolysis and/or endovascular therapy will be prospectively enrolled.

At intervention sites, clinicians may use the LingBao System during their routine workflows. The platform integrates routinely available clinical and imaging data, automatically estimates onset-to-treatment windows, screens contraindications, and provides evidence-based, guideline-concordant recommendations for reperfusion therapy; all treatment decisions remain at physician discretion.

The primary endpoint is the 90-day modified Rankin Scale (mRS) score analyzed by ordinal shift. Secondary endpoints include workflow metrics (door-to-needle time and door-to-puncture time), reperfusion treatment rates, early neurological improvement, symptomatic intracranial hemorrhage, and mortality.

The study plans to include approximately 20 centers (about 150 patients per center), accounting for intracluster correlation. The findings will provide real-world evidence on the clinical value of AI-assisted decision support for reperfusion therapy in AIS and inform broader implementation of intelligent stroke management systems.

DETAILED DESCRIPTION:
The LingBao System (Stroke Reperfusion Intelligent Decision System, SRIDS) is an AI-based clinical decision support platform designed to assist physicians in the evaluation and treatment decision-making process for acute ischemic stroke (AIS) patients eligible for reperfusion therapy. Built upon the 2024 Chinese Guidelines for Reperfusion Therapy in Acute Ischemic Stroke, major international randomized controlled trial (RCT) evidence, and large-scale real-world datasets, LingBao integrates clinical information, imaging parameters, and guideline-based criteria to provide transparent, evidence-graded recommendations for intravenous thrombolysis and/or endovascular therapy.

This multicenter, cluster-randomized controlled trial aims to assess the real-world effectiveness and safety of LingBao in optimizing reperfusion decision-making and improving patient outcomes. Twenty certified stroke centers in China will be randomized 1:1 to either LingBao-assisted care or standard care. Consecutive adult patients (≥18 years) presenting within 24 hours of last-known-well and evaluated for reperfusion therapy will be prospectively enrolled.

At intervention sites, clinicians may use LingBao during standard clinical workflows. The system automatically calculates the estimated onset-to-treatment window, screens contraindications, summarizes imaging-based eligibility criteria, and displays guideline-concordant recommendations along with their class and level of evidence. LingBao does not replace physician judgment; all clinical decisions remain entirely at the discretion of the treating team.

Data on patient demographics, baseline characteristics, workflow times, treatments, and outcomes will be collected through standardized electronic case report forms (eCRFs). The primary outcome is functional status at 90 days, measured by the modified Rankin Scale (mRS) and analyzed using an ordinal shift model. Key secondary outcomes include door-to-needle time (DNT) for intravenous thrombolysis, door-to-puncture time (DPT) for endovascular therapy, rates of reperfusion treatment, early neurological improvement, symptomatic intracranial hemorrhage, and mortality.

By systematically integrating AI-driven clinical reasoning with evidence-based medicine, the LingBao study aims to establish an intelligent, reproducible, and guideline-concordant framework for acute stroke management. The results are expected to inform large-scale implementation of AI-supported decision systems to enhance the quality, consistency, and efficiency of stroke reperfusion therapy in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Clinical diagnosis of acute ischemic stroke (AIS).
* Presentation within 24 hours of symptom onset or last-known-well.
* Evaluated for reperfusion therapy (intravenous thrombolysis and/or endovascular treatment).
* Admission to one of the participating certified stroke centers.
* Availability of required clinical and imaging data for system evaluation and outcome assessment.

Exclusion Criteria:

* Absence of key clinical or imaging data necessary for analysis.
* Patients not undergoing reperfusion assessment or outside the pre-defined workflow.
* Prior participation in LingBao pilot testing or other AI-based decision support trials within the past 6 months.
* Explicit refusal of data use or withdrawal of consent (if applicable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Functional outcome at 90 days assessed by the modified Rankin Scale (mRS) | 90 days post-stroke onset
  Functional status at 90 days after stroke onset will be measured using the modified Rankin Scale (mRS, range 0-6). Outcomes will be analyzed as an ordinal shift across the full mRS distribution, comparing LingBao-assisted care versus standard care.

SECONDARY OUTCOMES:
Door-to-Needle Time (DNT) for Intravenous Thrombolysis at baseline | Baseline
  Time interval between hospital arrival and initiation of intravenous thrombolysis among patients receiving IVT.
Door-to-Puncture Time (DPT) for Endovascular Therapy at baseline | Baseline
  Time interval between hospital arrival and arterial puncture for patients undergoing endovascular therapy.
Reperfusion Treatment Rate at baseline | Baseline
  Proportion of eligible acute ischemic stroke patients who received intravenous thrombolysis and/or endovascular therapy.
Symptomatic Intracranial Hemorrhage (sICH) within 36 hours after treatment | Within 36 hours after treatment
  Occurrence of symptomatic intracranial hemorrhage within 36 hours after reperfusion therapy, defined according to ECASS III criteria.
All-Cause Mortality at 90 days post-stroke onset | 90 days post-stroke onset
  All-cause mortality within 90 days after stroke onset.